CLINICAL TRIAL: NCT02732275
Title: A Phase 1 Multiple Ascending Dose Study of DS-3201b in Subjects With Lymphomas
Brief Title: DS-3201b in Participants With Lymphomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-A-J101; 163173 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma, Malignant; Non-hodgkin Lymphoma
Keywords: Adult T-cell leukemia-lymphoma (ATL); Peripheral T-cell lymphoma (PTCL); Cutaneous T-cell lymphoma (CTCL); B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Leukemia-Lymphoma, Adult T-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation - DS-3201b (Experimental): Dose escalation is to identify the recommended phase 2 dose of DS-3201b guided by the modified continuous reassessment method using a Bayesian logistic regression model following escalation.
  Interventions: Drug: DS-3201b
- Dose Expansion - DS-3201b (Experimental): Part 2 is a dose expansion to examine the safety and efficacy of DS-3201b.
  Interventions: Drug: DS-3201b

INTERVENTIONS:
Drug: DS-3201b — DS-3201 to be administered orally once daily in each 28-day cycle.
  Arms: Dose Escalation - DS-3201b
Drug: DS-3201b — DS-3201 to be administered orally once daily in each 28-day cycle at the recommended dose for expansion.
  Arms: Dose Expansion - DS-3201b

SUMMARY:
DS-3201b is an experimental drug that is being investigated in clinical research.

Adults with non-Hodgkin lymphoma (NHL) may be able to join this study if their disease has come back after remission or is not responding to current treatment

This study has three parts. The Dose Escalation part is designed is to find the safe dose of DS-3201b that adults with advanced NHL can tolerate. The Dose Expansion phase will determine how effective DS-3201b is for rare types of NH and collect additional safety data. Last, the Drug-Drug Interaction (DDI) Cohort (US Only) will evaluate the effect of DS-3201b on the pharmacokinetics (PK) of midazolam and digoxin when co-administered to patients with NHL

ELIGIBILITY:
Inclusion Criteria:

* Has hematocytological or pathological diagnosis of non- Hodgkin's lymphoma (NHL)
* Has relapsed from or is refractory to standard treatment or no standard treatment is available
* Is the age of majority in their country (18 in the US and 20 in Japan) at the time of informed consent
* Has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Has at least one evaluable lesion site (not applicable for the DDI cohort)
* Has preserved organ function based on baseline laboratory data at screening tests
* If of reproductive potential, agrees to avoid harvesting ova or sperm, and to use a protocol-defined form of contraception or avoid intercourse, during and upon completion of the study, and for at least 3 months after the last dose of study drug
* Tumor biopsy collections:

  1. willing to provide archived or fresh tumor tissue samples that are sufficient for comprehensive genomic and/or proteomic analyses at baseline
  2. [US only] willing to provide fresh on-treatment tumor biopsy if deemed acceptable risk by the investigator

     [Japan only] fresh on-treatment tumor biopsy should be performed if deemed acceptable risk by the investigator
  3. willing to provide optional fresh end-of-treatment biopsy

For ATL subjects:

* Has a positive test result for human T-lymphotropic virus type I antibody
* Has ATL subtype classified as acute, lymphomatous, or chronic with poor prognostic factor
* Has diagnosis of relapse (including relapse after partial remission [PR]) or treatment-resistant ATL at the time of informed consent after prior treatment with at least 1 anti-cancer medication regimen

Exclusion Criteria:

* Has been diagnosed with protocol-defined cutaneous T-cell lymphoma or T-cell leukemia. For DDI cohort, CTCL is not exclusionary.
* Has a history or presence of central nervous system (CNS) involvement
* Has a medical history, complication or other malignancy considered inappropriate for participation in the study, or a serious physical or psychiatric disease, the risk of which may be increased by participation in the study
* Has received drugs or other treatments not allowed by the protocol
* History of treatment with other enhancer of zeste (EZH) inhibitors
* Has had allogeneic hematopoietic stem cell transplantation (HTCP) within 90 days before scheduled dosing on Cycle 1 Day 1
* Is pregnant or breastfeeding
* Is otherwise deemed ineligible to participate by the investigator or sub-investigator

DDI Cohort Only:

* Has received following medications within 14 days prior to study drug administration
* Any CYP3A inhibitors/inducers including weak CYP3A inhibitors/inducers, and P-gp inhibitors, midazolam as well as digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Period: Number of participants with dose-limiting toxicities (DLTs) | within 28 days after the initial dose of the study drug
  Number of DLT-evaluable participants with protocol-defined DLTs
Dose Escalation Period: Maximum concentration (Cmax) of DS-3201 | within the first 28-day cycle
  Categories: Cycle 1 Day 1, Cycle 1 Day 15
Dose Escalation Period: Time of maximum concentration (Tmax) of DS-3201 | within the first 28-day cycle
  Categories: Cycle 1 Day 1, Cycle 1 Day 15
Dose Escalation Period: Area under the plasma concentration time curve up to the last quantifiable time (AUClast) for DS-3201 | Day 1 of the first 28-day cycle
Dose Escalation Period: Area under the plasma concentration time curve during the dosing interval (AUCtau) for DS-3201 | Day 1 of the first 28-day cycle
Dose Escalation Period: Trough (minimum) plasma concentration (Ctrough) | Day 15 of the first 28-day cycle
Dose Escalation Period: Average plasma concentration (Cavg) | Day 15 of the first 28-day cycle
DDI cohort only: Maximum concentration (Cmax) of DS-3201, midazolam, digoxin | within the first 28-day cycle
  Categories: Day -4, Cycle 1 Day 1, Cycle 1 Day 15
DDI cohort only: Time of maximum concentration (Tmax) of DS-3201, midazolam, digoxin | within the first 28-day cycle
  Categories: Day -4, Day 0 (for alternate schedule), Cycle 1 Day 1, Cycle 1 Day 15
DDI cohort only: Area under the plasma concentration time curve up to the last quantifiable time (AUClast) for DS-3201,midazolam,digoxin | within the first 28-day cycle
  Categories: Day -4, Day 0 (for alternate schedule), Cycle 1 Day 1, Cycle 1 Day 15
DDI cohort only: Area under the plasma concentration time curve during the dosing interval (AUCtau) for DS-3201, midazolam, digoxin | within the first 28-day cycle
  Cycle 1 Day 1, Cycle 1 Day 15
Number of participants with treatment-emergent adverse events (TEAEs) | through the end of the study (within approximately 5 years)
  TEAEs are systematically collected from lab values, physical exams, and other investigations

SECONDARY OUTCOMES:
Best overall response, based on international consensus criteria | from the start of study treatment to the end of follow-up visit (within 5 years)
  Best overall response is defined as the percentage of participants who achieved each category as the best response, considering all overall responses assessed at all time points after the start of study treatment.
  Categories: CR, CRu, PR, SD, RD/PD, UA
  Categories: Malignant lymphoma, ATL, CTCL
Objective response rate (ORR) | within 5 years
  ORR is defined as the percentage of participants who were assessed for best overall response, who achieved CR, CRu, or PR
Disease control rate (DCR) | within 5 years
  DCR is defined as the percentage of participants who were assessed for best overall response, who achieved a best response of CR, CRu, PR, or SD
Duration of response (DOR) | within 5 years
  DOR is defined as the time from the date at which criteria are first met for CR or PR (including CRu for ATL) until the first date that progressive disease is objectively documented.
Progression-free survival (PFS) | witihn 5 years
  PFS is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of disease progression or death due to any cause.
Number of participants with malignant lymphoma who achieved each level of therapeutic response per international consensus standards | through the end of the study (within approximately 5 years)
  Categories: Complete remission (CR), Partial remission (PR), Stable disease (SD), Relapsed disease or progressive disease (RD/PD)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, MD, Study Director — Daiichi Sankyo
Locations (20):
- United States (10):
  - City of Hope National Medical center, Duarte, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center and James Cancer Hospital, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Japan (10):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kahiwa-shi, Chiba
  - Iwate Medical University Hospital, Morioka, Iwate
  - Imamura General Hospital, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Kumamoto University Hosipital, Kumamoto, Kumamoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - The Institute of Medical Science, The University of Tokyo, Minato-ku, Tokyo
  - National Cancer Center Hospital, Chūōku, Toyko

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Maruyama D, Jacobsen E, Porcu P, Allen P, Ishitsuka K, Kusumoto S, Narita T, Tobinai K, Foss F, Tsukasaki K, Feldman T, Imaizumi Y, Izutsu K, Morishima S, Yamauchi N, Yuda J, Brammer JE, Kawamata T, Ruan J, Nosaka K, Utsunomiya A, Wang J, Zain J, Kakurai Y, Yamauchi H, Hizukuri Y, Biserna N, Tachibana M, Inoue A, Horwitz SM. Valemetostat monotherapy in patients with relapsed or refractory non-Hodgkin lymphoma: a first-in-human, multicentre, open-label, single-arm, phase 1 study. Lancet Oncol. 2024 Dec;25(12):1589-1601. doi: 10.1016/S1470-2045(24)00502-3. Epub 2024 Oct 29. PMID 39486432